CLINICAL TRIAL: NCT01216033
Title: An Exploratory Study to Evaluate the Distribution of [111In]ABY-025 Uptake for SPECT Imaging in Subjects With Metastatic Breast Cancer
Brief Title: Exploratory Study of Breast Cancer With ABY025
Acronym: ABY0125
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biomedical Radiation Sciences (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Dr. Henrik Lindman, Uppsala Akademiska Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 111InABY025
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Diagnostics; HER2; Imaging; Metastases; SPECT; Imaging of metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 111-In-ABY-025 — Intravenous injection of the agent

SUMMARY:
The aim is to study if breast cancer metastases accumulate the newly developed HER2 binding molecule 111-In-ABY025 and if that shows whether the metastases express HER2.

ELIGIBILITY:
Inclusion Criteria:

* female age >20 years
* one or more known metastases localizations

Exclusion Criteria:

* other critical disease than breast cancer
* age ≤ 20 years

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Imaging of metastases | One year
  Imaging of breast cancer metastases using 111-In-ABY015 for SPECT

SECONDARY OUTCOMES:
Can the new molecule be used for imaging in extended studies | October 2010 - June 2011

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska Hospital, Uppsala, Uppland, Sweden

REFERENCES:
- [Background] Carlsson J, Nordgren H, Sjostrom J, Wester K, Villman K, Bengtsson NO, Ostenstad B, Lundqvist H, Blomqvist C. HER2 expression in breast cancer primary tumours and corresponding metastases. Original data and literature review. Br J Cancer. 2004 Jun 14;90(12):2344-8. doi: 10.1038/sj.bjc.6601881. PMID 15150568